CLINICAL TRIAL: NCT03627728
Title: Phase II Randomized Study of Maintenance Regorafenib vs Placebo in no Progression Patients After First-line Platinum and Fluoropyrimidines Based Chemotherapy in HER2 Negative Locally Advanced/Metastatic Gastric or Gastroesophagel Junction Cancer (a-MANTRA Study)
Brief Title: Study Maintenance Regorafenib vs Placebo, no Progression Patients After I Line Chemotherapy Metastatic Gastric Cancer
Acronym: a-MANTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOIRC-05-2016
Record Dates: First submitted 2018-05-18; First posted 2018-08-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- regorafenib (Experimental): Regorafenib 160 mg, 4 tablets once daily on days 1-21, every 4 weeks, until intolerance or progression disease
  Interventions: Drug: Regorafenib
- placebo (Placebo Comparator): Placebo 4 tablets once daily on day 1-21, every 4 weeks, until intolerance or progression disease
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Regorafenib — regorafenib/placebo
  Other Names: stivarga
  Arms: regorafenib
Other: placebo — regorafenib/placebo
  Arms: placebo

SUMMARY:
Randomized, double-blind, placebo-controlled, multicenter Phase-II study.

Approximately 120 subjects with CR/PR/SD after platinum compounds and fluoropyrimidines based regimens: up to 6 cycles of cisplatin and 5-fluorouracil or capecitabine, up to 12 cycles of FOLFOX, up to 8 cycles of XELOX, will be randomly assigned (1:1 ratio) to one of the following treatment groups:

Arm A: Placebo 4 tablets once daily on day 1-21, every 4 weeks, until intolerance or progression disease Arm B: Regorafenib 160 mg, 4 tablets once daily on days 1-21, every 4 weeks, until intolerance or progression disease Primary Variable: PFS1

ELIGIBILITY:
Inclusion Criteria:

1. Male of female ≥ 18 years of age
2. Have an Eastern Cooperative Oncology Group performance status of 0 or 1 within 14 days prior to the initiation of study treatment
3. Diagnosis of histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction
4. HER2 negative gastric or gastroesophagel junction cancer ( ICH 0, IHC 1+, IHC + FISH -)
5. Locally advanced/metastatic gastric or gastroesophageal junction cancer
6. CR/PR/SD after first-line platinum compound and Fluoropyrimidines based chemotherapy
7. Measurable disease according to RECIST 1.1 criteria
8. Have adequate bone marrow function, liver function, and renal function, as measured by the following laboratory assessments conducted within 7 days prior to the initiation of study treatment:
9. Total bilirubin 1.5 times the upper limit of normal (ULN)
10. Alanine aminotransferase and aspartate aminotransferase 3 times the ULN
11. Lipase 1.5 times the ULN
12. Serum creatinine 1.5 times the ULN
13. Glomerular filtration rate 30 mL/min/1,73 m2 according to the Modified Diet in Renal Disease abbreviated formula
14. International normalized ratio of prothrombin time and activated partial thromboplastin time 1.5 times the ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate if no underlying abnormality in coagulation parameters exists per medical history.
15. Platelet count 100,000 /mm3, hemoglobin 9 g/dL, absolute neutrophil count 1500/mm3 without transfusions or granulocyte colony stimulating factor and other hematopoietic growth factors
16. Alkaline phosphatase ≤ 2.5 times the ULN
17. Understand, be willing to give consent, and sign the written informed consent form (ICF) prior to undergoing any study-specific procedure.
18. If female and of childbearing potential, have a negative result on a pregnancy test performed a maximum of 7 days before initiation of study treatment.
19. If female and of childbearing potential, or if male, agree to use adequate contraception (eg, abstinence, intrauterine device, oral contraceptive, or double-barrier method) based on the judgment of the investigator or a designated associate from the date on which the ICF is signed until 8 weeks after the last dose of study drug.

Exclusion Criteria:

1. Are taking strong cytochrome P (CYP) CYP3A4 inhibitors (eg, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, voriconazole) or strong CYP3A4 inducers (eg, carbamazepine, phenobarbital, phenytoin, rifampin, St. John's Wort)
2. Have used biologic response modifiers, such as G-CSF, within 3 weeks of study entry
3. Have had prior treatment with regorafenib or any other VEGFR-targeting kinase inhibitor.
4. Completed their last dose of chemotherapy more than 8 weeks, whichever came later, prior to randomization.
5. Have had prior or concurrent cancer distinct in primary site or histology from GC or GJC within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, no-melanoma skin cancer, or superficial bladder tumors classified as noninvasive tumor (Ta), carcinoma in situ (Tis), or tumor invades lamina propria (T1).
6. Have had systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and/or hormonal therapy within 4 weeks prior to initiation of study treatment.
7. Have unresolved toxicity higher than National Cancer Institute-Common Terminology for Adverse Events version 4.0 (NCI-CTCAE v 4.0) Grade 1 attributed to any prior therapy/procedure, excluding alopecia and/or oxaliplatin-induced neurotoxicity ≤ Grade 2 and hemoglobin ≥ 9 g/dL as per inclusion criteria
8. Have had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment.
9. Are pregnant.
10. Are breastfeeding.
11. Are unable to swallow oral tablets (crushing of study treatment tablets is not allowed).
12. Have congestive heart failure classified as New York Heart Association Class 2 or higher
13. Have had unstable angina (angina symptoms at rest) or new-onset angina 3 months prior to screening.
14. Have had a myocardial infarction 6 months prior to initiation of study treatment.
15. Have cardiac arrhythmias requiring anti-arrhythmic therapy, with the exception of beta blockers or digoxin.
16. Have uncontrolled hypertension (systolic blood pressure [SBP] 140 mmHg or diastolic blood pressure [DBP] 90 mmHg) despite optimal medical management.
17. Have had arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within 6 months prior to the initiation of study treatment.
18. Have an ongoing infection with severity of Grade 2 or above (NCI-CTCAE v 4.0).
19. Have a known history of human immunodeficiency virus infection.
20. Have either active or chronic hepatitis B or C requiring treatment with antiviral therapy.
21. Have a seizure disorder requiring medication.
22. Have a history of organ allograft.
23. Have evidence or history of any bleeding diathesis (including mild hemophilia), irrespective of severity.
24. Have had a hemorrhage or a bleeding event Grade 3 (NCI-CTCAE v 4.0) within 4 weeks prior to the initiation of study treatment.
25. Have a nonhealing wound, ulcer, or bone fracture.
26. Have renal failure requiring hemodialysis or peritoneal dialysis.
27. Have dehydration Grade 1 (NCI-CTCAE v 4.0).
28. Have interstitial lung disease with ongoing signs and symptoms at the time informed consent is obtained.
29. Have persistent proteinuria > 3.5 g/24 hours measured by urine protein creatinine ratio from a random urine sample (Grade 3, NCI-CTCAE v 4.0).
30. Have any other serious or unstable illness, or medical, psychological, or social condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results.
31. Have a known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation of the study drugs.
32. Have any malabsorption condition.
33. Have a close affiliation with the investigational site (eg, be a close relative of the investigator) or be a dependent person (eg, be an employee or student working at the investigational site).
34. Untreated gastro-esophageus varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
PFS1 | 36 months
  Progression free survival will be calculated for all patients from the date of randomization until the date PD or death is first reported.

SECONDARY OUTCOMES:
OS | 36 months
  time from date of randomization to the date of Death from any cause
PFS2 | 36 months
  PFS 2 will be calculated from the start of second line therapy to PD or death
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability | 36 months
  The overall incidences of AEs will be summarized. Patients who experienced the same event on more than one occasion are counted only once in the calculation of the event frequency, at the highest intensity ever observed.
Response Rate | 36 months
  in patients who are randomized at enrollment to treatment with regorafenib vs placebo,
quality of life To compare the patient treatment-related symptoms | up to 8 months
  To compare the patient treatment-related symptoms as measured by the European Organization for research and treatment of cancer EORTC QLQ-C30, (days 1, week , 8, 16, 24, 32) , for patients in each treatment arm.
biomarker evaluation | 36 months
  To correlate the genetic mutational profile of the tumors with the RR and the OS of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Pinto, MD, Principal Investigator — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (1):
- Struttura Complessa di OncologiaIRCCS- Istituto in Tecnologie Avanzate e Modelli Assistenziali in Oncologia Arcispedale Santa Maria Nuova, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No